CLINICAL TRIAL: NCT02783638
Title: A Open-label, Randomized, Crossover Clinical Trial to Assess the PK of Pregabalin CR After Multiple Dosing as Compared to Pregabalin IR and the Food Effect of High Fat Diet After Single Dosing in Healthy Male Volunteers
Brief Title: PK and Food Effect of Pregabalin Study After Dosing in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHD1119-102
Record Dates: First submitted 2016-02-15; First posted 2016-05-26 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2016-11

CONDITIONS: Peripheral Neuropathy Pain
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- YHD1119 (Pregabalin 300mg) (Experimental): YHD1119 (Pregabalin 300mg)
  Interventions: Drug: YHD1119
- Lyrica (Pregabalin 150mg) (Active Comparator): Lyrica (Pregabalin 150mg)
  Interventions: Drug: Lyrica

INTERVENTIONS:
Drug: YHD1119 — 2 by 2
  Other Names: Pregabalin 300mg
  Arms: YHD1119 (Pregabalin 300mg)
Drug: Lyrica — 2 by 2
  Other Names: Pregabalin 150mg
  Arms: Lyrica (Pregabalin 150mg)

SUMMARY:
This study is to assess the pharmacokinetics of Pregabalin controlled release formulation after multiple dosing as compared to Pregabalin immediate release formulation and the food effect of high fat diet after single dosing in healthy male volunteers.

DETAILED DESCRIPTION:
Cohort 1 study is to assess the PK of Pregabalin controlled release formulation as compared to Pregabalin immediate release formulation. Cohort 1 subjects will be admitted to the clinic at Day 1. All subjects will receive multiple dosing for three days of YHD1119 or Pregabalin IR and will remain in the clinic until completion of all assessment on Day 19 including collection of PK sample. The treatment periods were separated by a washout period (10-17 days).

Cohort 2 study is to assess the food effect of high fat diet after single dosing. Cohort 2 subjects will be admitted to the clinic at Day -1. All subjects will receive a single dose of YHD1119 and will remain in the clinic until completion of all assessment on Day 9 including collection of PK sample. The treatment periods were separated by a washout period (7-14 days).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male with body mass index (BMI) between 18.5 and 28 kg/m2
* Who has not suffered from clinically significant disease
* Provision of signed written informed consent

Exclusion Criteria:

* History of and clinically significant disease
* A history of drug abuse or the presence of positive reactions to drugs that have abuse potential in urine screenings for drugs
* Administration of other investigational products within 3 months prior to the first dosing

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cohort 1: Cmax | Lyrica(Pregabalin 150mg): 0.33,0.67,1,2,4,8,12,12.33,12.67,13,14,16,20,24,36 hours
Cohort 1: AUCtau | Lyrica(Pregabalin 150mg): 0.33,0.67,1,2,4,8,12,12.33,12.67,13,14,16,20,24,36 hours
Cohort 1: Cmax | YHD1119(Pregabalin 300mg): 1,2,3,4,5,6,8,10,12,16,24,36 hours
Cohort 1: AUCtau | YHD1119(Pregabalin 300mg): 1,2,3,4,5,6,8,10,12,16,24,36 hours
Cohort 2: Cmax | YHD1119(Pregabalin 300mg): 1,2,3,4,5,6,8,10,12,16,24,36 hours
Cohort 2: AUCtau | YHD1119(Pregabalin 300mg): 1,2,3,4,5,6,8,10,12,16,24,36 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No